CLINICAL TRIAL: NCT00432562
Title: A Bioequivalence Study of Vinorelbine Tartrate Injectable Emulsion (ANX-530) in Patients With Advanced Cancer.
Brief Title: A Bioequivalence Study of Vinorelbine Tartrate Injectable Emulsion in Patients With Advanced Cancer.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mast Therapeutics, Inc. (Industry)
Collaborators: Synteract, Inc. (Industry); Thywill Latam Solutions SRL (Unknown); OCASA Soluciones Logísticas S.A. (Unknown); Worldwide Clinical Trials (Other)
Responsible Party: Chief Executive Officer, Adventrx Pharmaceuticals, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 530-01
Record Dates: First submitted 2007-02-06; First posted 2007-02-08 (Estimated); Results first posted 2012-02-23 (Estimated); Last update posted 2012-02-23 (Estimated); Status verified 2012-01

CONDITIONS: Breast Cancer; Non-small Cell Lung Cancer; Non-Hodgkins Lymphoma
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Lymphoma, Non-Hodgkin | interventions — Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Vinorelbine Tartrate — Subjects received one dose each of ANX-530 and NAVELBINE, each providing 30 mg/m2 vinorelbine. Study drugs will be infused into an arm vein over ten minutes.
  Other Names: Exelbine (proposed); ANX-530

SUMMARY:
This study was a randomized, single dose crossover comparison of the investigational product with a Reference Product (vinorelbine tartrate injection, NAVELBINE®). The primary objective was to demonstrate the equivalence of ANX-530 and the Reference Product, NAVELBINE.

DETAILED DESCRIPTION:
ANX-530 (vinorelbine tartrate injectable emulsion), an investigational drug, is an oil-in-water emulsion of vinorelbine tartrate composed of an oil phase and emulsifier dispersed in an aqueous solution. ADVENTRX Pharmaceuticals, Inc. of San Diego, California, developed ANX-530 as a vinorelbine tartrate formulation to be used in clinical settings where Vinorelbine Tartrate Injection (NAVELBINE) is indicated. Nonclinical toxicology studies suggest either equivalent or less toxicity of ANX-530 compared to Reference Product. In particular, ANX-530 caused less vein toxicity in a rabbit vein irritation model, suggesting ANX-530 could potentially cause less venous irritation than NAVELBINE in a clinical setting. ADVENTRX is investigating whether ANX-530 could substitute for NAVELBINE in these settings.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Advanced cancer potentially sensitive to vinorelbine:
* Breast cancer.
* Stage 3 or 4 non-small cell lung cancer.
* Non-Hodgkins lymphoma.
* Cancer of other histologic type, sensitive to vinca alkaloids.
* Rare tumor type with no standard treatment, for which single agent vinorelbine is appropriate therapy.
* Failure of standard treatment(s) of the tumor.
* Life expectancy of at least three months.
* ECOG performance level 0-2 or Karnofsky score 100-70.
* Hematological and serum chemistry results with defined ranges.
* Willingness and ability to provide written informed consent.

Exclusion Criteria:

* Pregnancy or lactation. In a woman of childbearing potential, a positive pregnancy test result, no pregnancy test result, or no use of reliable contraception, at baseline. A postmenopausal woman will be considered to be of childbearing potential until there has been amenorrhea for at least 12 consecutive months.
* Previous treatment with vinorelbine or mitomycin.
* Any history suggesting or demonstrating resistance to, lack of response to, or intolerance of any prior vinca alkaloid treatment.
* Active infection.
* Prior anticancer therapy completed within four weeks prior to the first day of study treatment.
* Failure to have recovered from any toxicity of previous cancer treatment (patients with alopecia will not be excluded).
* Participation in another experimental drug study within four weeks prior to the first day of study treatment.
* Requirement for any concomitant chemotherapeutic agent other than the study medication.
* Any investigator judgment that the individual would not be an appropriate study subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-02; Primary Completion 2007-11 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lino Arboit, M.D., Principal Investigator — Fundación Centro Oncológico de Integración Regional - COIR.; Gerardo F Arroyo, M.D., Principal Investigator — Hospital Privado De Santa Clara De Asis; Cesar R Blajman, M.D., Principal Investigator — Isis Clínica Especializada; Matias Chacon, M.D., Principal Investigator — Instituto Médico Espcializado Alexander Fleming; Luis E Fein, M.D., Principal Investigator — Centro Oncológico; Hugo R. Requejo, M.D., Principal Investigator — Hospital Regional De Concepción; Edgar P Quintana, M.D., Principal Investigator — CIMA Salud
Locations (5):
- Argentina (5):
  - Clinical Investigative Site, Buenos Aires
  - Clinical Investigative Site, Mendoza
  - Clinical Investigative Site, Rosario
  - Clinical Investigative Site, San Miguel de Tucumán
  - Clinical Investigative Site, Santa Fe

RESULTS

PARTICIPANT FLOW:
Recruitment Details: STUDIED PERIOD:
  First Patient Enrolled: 22 March 2007 Last Patient Completed: 02 November 2007 Study patients were enrolled at seven study sites in Argentina.
Pre-assignment Details: Pre-screening data was not collected for this study
Groups:
- ANX-530/Navelbine: Patients were randomly assigned to receive a single intravenous (IV) dose of 30 mg/m2 of ANX 530 in the first study period, then one week later patients crossed over to receive a single IV dose of 30 mg/m2 of Navelbine in the second study period.
- Navelbine/ANX-530: Patients were randomly assigned to receive a single intravenous (IV) dose of 30 mg/m2 of Navelbine in the first study period, then one week later patients crossed over to receive a single IV dose of 30 mg/m2 of ANX-530 in the second study period.
Period: Overall Study
Arm/Group | ANX-530/Navelbine | Navelbine/ANX-530
Started | 16 | 15
Completed | 13 | 15
Not Completed | 3 | 0
Not completed — Death | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ANX-530/Navelbine | Navelbine/ANX-530 | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 21
  >=65 years | 5 | 5 | 10
Age Continuous [Mean (Standard Deviation); unit: years] | 62.2 (12.77) | 58.0 (13.34) | 60.2 (13.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Male | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  Argentina | 16 | 15 | 31

OUTCOME MEASURES:

1. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: 0-144 hours post dose
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ANX-530 | Navelbine
Number analyzed (Participants) | 31 | 31
hours | 0.35 (0.13) | 0.34 (0.08)

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: 0-144 hours post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ANX-530 | Navelbine
Number analyzed (Participants) | 31 | 31
ng/mL | 227 (108) | 223 (125)

3. Primary Outcome: Area Under the Plasma Concentratio-Time Curve From Time 0 to the Time of the Last Measurable Concentration (AUClast)
Description: Determined Using the Linear Trapezoidal Rule
Time Frame: 0-144 hours post-dose
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | ANX-530 | Navelbine
Number analyzed (Participants) | 31 | 31
hr*ng/mL | 757.8 (363.7) | 716.1 (272.6)

4. Primary Outcome: Area Under the Concentration-Time Curve From Time 0 to Infinity (AUCinf)
Description: AUCinf = AUClast + (Clast/lamda z)
Time Frame: 0-144 hours post-dose
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | ANX-530 | Navelbine
Number analyzed (Participants) | 31 | 30
hr*ng/mL | 810.1 (400.9) | 718.5 (223.5)

5. Primary Outcome: Percentage of AUCinf Based on Extrapolation (AUCextrap)
Time Frame: 0-144 hours post-dose
Measure: Mean (Standard Deviation); unit: % of participants
Arm/Group | ANX-530 | Navelbine
Number analyzed (Participants) | 31 | 30
% of participants | 6.23 (2.54) | 4.72 (3.11)

6. Primary Outcome: Observed Elimination Rate Constant Associated With the Terminal Portion of the Curve (λ z)
Description: Estimated via linear regression of the time versus log concentration
Time Frame: 0-144 hours post-dose
Measure: Mean (Standard Deviation); unit: hr-1
Arm/Group | ANX-530 | Navelbine
Number analyzed (Participants) | 31 | 30
hr-1 | 0.0160 (0.0044) | 0.0187 (0.0062)

7. Primary Outcome: Observed Terminal Elimination Half-Life (t1/2)
Description: t1/2 = [ln(2)/λ z]
Time Frame: 0-144 hours post-dose
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ANX-530 | Navelbine
Number analyzed (Participants) | 31 | 30
hours | 46.50 (12.43) | 40.48 (13.50)

8. Primary Outcome: Time of Last Measurable Concentration (Tlast)
Time Frame: 0-144 hours post-dose
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ANX-530 | Navelbine
Number analyzed (Participants) | 31 | 31
hours | 141.83 (12.93) | 141.79 (12.92)

9. Primary Outcome: Last Quantifiable Drug Concentration (Clast)
Time Frame: 0-144 hours post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ANX-530 | Navelbine
Number analyzed (Participants) | 31 | 31
ng/mL | 0.819 (0.834) | 0.824 (1.31)

10. Primary Outcome: Mean Residence Time (MRTinf)
Description: MRT = (AUMCinf)/(AUCinf)
Time Frame: 0-144 hours post-dose
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ANX-530 | Navelbine
Number analyzed (Participants) | 31 | 30
hours | 35.39 (7.90) | 31.31 (10.06)

ADVERSE EVENTS:
Time Frame: AEs and their treatment were documented from the time of the first dose of study medication until 30 days after the last dose. Mild, moderate and severe AEs not related to study treatment were followed for approx 30 days after the last study drug dose.
Description: Events that were serious, life threatening or related to study treatment were followed until resolution, downgrading of an SAE to non-serious, subject death, start of new cancer therapy or re-assessment of the event's relationship to study medication.
Groups:
- ANX-530/Navelbine: Patients were randomly assigned to receive a single intravenous (IV) dose of 30 mg/m2 of ANX 530 in the first study period, then one week later patients crossed over to receive a single IV dose of 30 mg/m2 of Navelbine. Serious Adverse Events are reported by treatment-sequence group and not by study therapy group.
- Navelbine/ANX-530: Patients were randomly assigned to receive a single intravenous (IV) dose of 30 mg/m2 of Navelbine in the first study period, then one week later patients crossed over to receive a single IV dose of 30 mg/m2 of ANX-530. Serious Adverse Events are reported by treatment-sequence group and not by study therapy group.
Arm/Group | ANX-530/Navelbine | Navelbine/ANX-530
Serious Adverse Events (participants affected / at risk) | 5/16 | 1/15
Other Adverse Events (participants affected / at risk) | 21/31 | 22/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ANX-530/Navelbine (N=16) | Navelbine/ANX-530 (N=15)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
FEBRILE INFECTION (Infections and infestations) | 1 | 1
GENITAL INFECTION FEMALE (Infections and infestations) | 1 | 0
LEUKOPENIA (Blood and lymphatic system disorders) | 1 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 3 | 0
PNEUMONIA (Infections and infestations) | 1 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0
STUPOR (Nervous system disorders) | 1 | 0
COMA (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ANX-530/Navelbine (N=31) | Navelbine/ANX-530 (N=31)
ABDOMINAL PAIN (Gastrointestinal disorders) | 4 | 0
ANAEMIA (Blood and lymphatic system disorders) | 3 | 3
ASTHENIA (General disorders) | 3 | 2
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
CONSTIPATION (Gastrointestinal disorders) | 5 | 5
INFUSION SITE PHLEBITIS (General disorders) | 1 | 7
LEUKOPENIA (Blood and lymphatic system disorders) | 6 | 3
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0
NAUSEA (Gastrointestinal disorders) | 5 | 4
NEUTROPENIA (Blood and lymphatic system disorders) | 12 | 7
RASH (Skin and subcutaneous tissue disorders) | 3 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 2
VOMITING (Gastrointestinal disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of data related to the Study, including publication in special medical magazines, or the disclosure at medical congresses shall be previously authorized in writing by the Sponsor, whereby the Principal Investigator should present the material with an anticipation of not less than 60 days as from the publication or medical congress. The Sponsor decides upon the authorship of any publication related to the Study.